CLINICAL TRIAL: NCT05247489
Title: A Safety and Efficacy Study of Ruxolitinib Cream Combined With Narrow-Band Ultraviolet B Phototherapy in Participants With Vitiligo
Brief Title: A Study to Evaluate the Safety and Efficacy of Ruxolitinib Cream With Phototherapy in Participants With Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-217
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Vitiligo
Keywords: Non-segmental; Vitiligo; hypopigmentation; Pigment Disorders; Skin Diseases; JAK inhibitor
MeSH Terms: conditions — Vitiligo; Hypopigmentation; Pigmentation Disorders; Skin Diseases | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Ruxolitinib + Narrow-Band Ultraviolet B Phototherapy (NB-UVB) (Experimental): Participants will initially apply ruxolitinib 1.5%mg cream as a monotherapy. At week 12, those who have < 25% improvement in total body Vitiligo Area Scoring Index (T-VASI25) will have NB-UVB phototherapy added to their ruxolitinib 1.5% cream BID regimen. NB-UVB will be given 3 times per week starting at Week 12 through Week 48 (36 weeks). For participants who receive combination therapy, NB-UVB machines will be supplied by the sponsor for at home use during the study.
  Interventions: Drug: Ruxolitinib 1.5% cream; Device: NB-UVB phototherapy
- Group B: Ruxolitinib Monotherapy (Experimental): Participants will apply ruxolitinib 1.5% cream BID as monotherapy. Participants who have ≥ T-VASI25 at Week 12 will continue on ruxolitinib 1.5% cream BID alone.
  Interventions: Drug: Ruxolitinib 1.5% cream

INTERVENTIONS:
Drug: Ruxolitinib 1.5% cream — Ruxolitinib cream 1.5% applied twice a day (BID).
Device: NB-UVB phototherapy — NB-UVB (311-312 nm) phototherapy is an established treatment modality for vitiligo. Starting dose will be 200 mJ/cm2 and dose may be increased by 10% at each visit
  Other Names: Narrow-Band Ultraviolet B Phototherapy
  Arms: Group A: Ruxolitinib + Narrow-Band Ultraviolet B Phototherapy (NB-UVB)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ruxolitinib cream with or without phototherapy in adolescent and adult participants with non-segmental vitiligo for whom vitiligo area (facial and nonfacial) does not exceed 10% body surface area (BSA).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of nonsegmental vitiligo with depigmented area including all of the following:

  1. ≥ 0.5 F-VASI on the face
  2. ≥ 3.0 T-VASI (body areas not including the face)
  3. Total body vitiligo area (facial and nonfacial) not exceeding 10% BSA.
* Agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit. Over-the-counter preparations deemed acceptable by the investigator and camouflage makeups are permitted.

Exclusion Criteria:

* No pigmented hair within any of the vitiligo areas on the face.
* Other forms of vitiligo (eg, segmental) or other differential diagnosis of vitiligo or other skin depigmentation disorders.
* Used depigmentation treatments (eg, monobenzone) for past treatment of vitiligo or other pigmented areas.
* Previous adverse reaction to NB-UVB phototherapy that caused discontinuation of therapy.
* Lack of response (little or no repigmentation) to prior NB-UVB phototherapy.
* History of thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, ischemic stroke, myocardial infarction).
* Any other skin disease that, in the opinion of the investigator, would interfere with the study cream application or study assessments.
* Active acute bacterial, fungal, or viral skin infection (eg, herpes simplex, herpes zoster, chicken pox) within 1 week before baseline.
* Any serious illness or medical, physical, or psychiatric condition(s) that pose a significant risk to the participant; or interfere with interpretation of study data.
* Recent use of topical or systemic medications (including biologics or JAK inhibitors), or laser or phototherapy to treat vitiligo. Note: Recent may be defined differently for different treatments.
* Specific protocol-defined chemistry, hematology, and serological lab values.
* Those who are pregnant, lactating or considering pregnancy during the period of study participation.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, Study Director — Incyte Corporation
Locations (13):
- United States (11):
  - First Oc Dermatology, Fountain Valley, California
  - UC Davis Health, Sacramento, California
  - Palo Alto Medical Foundation, Sunnyvale, California
  - Delricht Clinical Research - Clinedge - Ppds Baton Rouge, Baton Rouge, Louisiana
  - Aesthetic and Dermatology Center, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Austin Institute For Clinical Research Aicr Pflugerville, Pflugerville, Texas
  - Principle Research Solutions, Spokane, Washington
- Canada (2):
  - Simcomed Health Ltd, Barrie, Ontario
  - Lynderm Research Inc, Markham, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 10 study centers in Canada and the United States.
Groups:
- Ruxolitinib 1.5% Cream BID: Participants who achieved ≥25% improvement in Total Body Vitiligo Scoring Index (T-VASI25) at Week 12 applied ruxolitinib 1.5% cream twice daily (BID) as monotherapy through Week 48.
- Ruxolitinib 1.5% Cream BID + NB-UVB: Participants applied ruxolitinib 1.5% cream BID as monotherapy through Week 12. Participants did not achieve T-VASI25 at Week 12 and added narrow-band ultraviolet B (NB-UVB) phototherapy to their ruxolitinib 1.5% cream BID regimen. NB-UVB phototherapy was given 3 times per week through Week 48 (up to 36 weeks). Participants continued to receive ruxolitinib 1.5% cream BID through Week 48.
Period: Overall Study
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Started | 20 | 35
Completed | 6 | 26
Not Completed | 14 | 9
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Withdrawn by Sponsor: Noncompliance | 0 | 1
Not completed — Left Country | 1 | 0
Not completed — Noncompliance with Investigational Product | 1 | 0
Not completed — Withdrawn by Sponsor: Surgery to Remove Excess Skin | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB | Total
Number analyzed (Participants) | 20 | 35 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (18.97) | 52.5 (14.25) | 48.7 (16.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 10 | 18 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 32 | 50
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 11 | 25 | 36
  Black/African-American | 1 | 2 | 3
  Asian | 6 | 6 | 12
  American-Indian/Alaska Native | 2 | 0 | 2
  East Indian | 0 | 1 | 1
  Arab | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Body Vitiligo Area Scoring Index (T-VASI) at Week 48
Description: T-VASI was calculated with contributions from 6 body sites. The percentage of vitiligo involvement was estimated in hand units (percentage of body surface area [BSA] estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each body site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; Week 48
Population: Full Analysis Set: all participants enrolled in the study who applied study cream at least once. Only participants with available data were analyzed. Change from Baseline was calculated as the Week 48 value minus the Baseline value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
scores on a scale
  Baseline | 6.58 (2.163) | 6.87 (2.103)
  Change from Baseline at Week 48: number analyzed (Participants) | 6 | 26
  Change from Baseline at Week 48 | -3.43 (1.219) | -3.46 (2.106)

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: up to approximately 52 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
Participants | 9 | 21

3. Secondary Outcome: Percentage of Participants Achieving a ≥50% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI50) Score at Each Post-Baseline Visit
Description: An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of participants
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | 6.3 [0.2 to 30.2] | 5.7 [0.7 to 19.2]
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | 21.4 [4.7 to 50.8] | 17.1 [6.6 to 33.6]
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | 63.6 [30.8 to 89.1] | 31.4 [16.9 to 49.3]
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | 85.7 [42.1 to 99.6] | 45.7 [28.8 to 63.4]
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | 100.0 [59.0 to 100.0] | 76.5 [58.8 to 89.3]
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | 100.0 [54.1 to 100.0] | 87.5 [71.0 to 96.5]
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | 100.0 [54.1 to 100.0] | 92.9 [76.5 to 99.1]
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | 100.0 [54.1 to 100.0] | 96.2 [80.4 to 99.9]

4. Secondary Outcome: Percentage of Participants Achieving a ≥75% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI75) Score at Each Post-Baseline Visit
Description: An F-VASI75 responder achieved at least 75% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of participants
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 10.0]
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | 45.5 [16.7 to 76.6] | 14.3 [4.8 to 30.3]
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | 57.1 [18.4 to 90.1] | 20.0 [8.4 to 36.9]
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | 85.7 [42.1 to 99.6] | 47.1 [29.8 to 64.9]
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | 83.3 [35.9 to 99.6] | 59.4 [40.6 to 76.3]
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | 100.0 [54.1 to 100.0] | 71.4 [51.3 to 86.8]
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | 100.0 [54.1 to 100.0] | 84.6 [65.1 to 95.6]

5. Secondary Outcome: Percentage of Participants Achieving a ≥90% Improvement From Baseline in the Face Vitiligo Area Scoring Index (F-VASI90) Score at Each Post-Baseline Visit
Description: An F-VASI90 responder achieved at least 90% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of participants
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 10.0]
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | 9.1 [0.2 to 41.3] | 0.0 [0.0 to 10.0]
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | 42.9 [9.9 to 81.6] | 2.9 [0.1 to 14.9]
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | 42.9 [9.9 to 81.6] | 17.6 [6.8 to 34.5]
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | 50.0 [11.8 to 88.2] | 34.4 [18.6 to 53.2]
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | 50.0 [11.8 to 88.2] | 53.6 [33.9 to 72.5]
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | 66.7 [22.3 to 95.7] | 53.8 [33.4 to 73.4]

6. Secondary Outcome: Percentage of Participants Achieving a ≥50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) Score at Each Post-Baseline Visit
Description: A T-VASI50 responder achieved ≥50% improvement from Baseline in T-VASI, calculated with contributions from 6 body sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to the nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each body site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of participants
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 10.0]
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | 18.2 [2.3 to 51.8] | 0.0 [0.0 to 10.0]
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | 42.9 [9.9 to 81.6] | 2.9 [0.1 to 14.9]
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | 71.4 [29.0 to 96.3] | 23.5 [10.7 to 41.2]
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | 66.7 [22.3 to 95.7] | 34.4 [18.6 to 53.2]
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | 83.3 [35.9 to 99.6] | 46.4 [27.5 to 66.1]
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | 83.3 [35.9 to 99.6] | 57.7 [36.9 to 76.6]

7. Secondary Outcome: Percentage of Participants Achieving a ≥75% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI75) Score at Each Post-Baseline Visit
Description: A T-VASI75 responder achieved ≥75% improvement from Baseline in T-VASI, calculated with contributions from 6 body sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to the nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each body site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of participants
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 10.0]
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 10.0]
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 10.0]
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | 28.6 [3.7 to 71.0] | 5.9 [0.7 to 19.7]
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | 50.0 [11.8 to 88.2] | 6.3 [0.8 to 20.8]
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | 50.0 [11.8 to 88.2] | 7.1 [0.9 to 23.5]
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | 50.0 [11.8 to 88.2] | 19.2 [6.6 to 39.4]

8. Secondary Outcome: Percentage of Participants Achieving a ≥90% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI90) Score at Each Post-Baseline Visit
Description: A T-VASI90 responder achieved ≥90% improvement from Baseline in T-VASI, calculated with contributions from 6 body sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to the nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each body site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of participants
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 10.0]
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 10.0]
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 10.0]
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 10.0]
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | 14.3 [0.4 to 57.9] | 2.9 [0.1 to 15.3]
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | 16.7 [0.4 to 64.1] | 3.1 [0.1 to 16.2]
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | 16.7 [0.4 to 64.1] | 7.1 [0.9 to 23.5]
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | 16.7 [0.4 to 64.1] | 7.7 [0.9 to 25.1]

9. Secondary Outcome: Change From Baseline in F-VASI at Each Post-Baseline Visit
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
scores on a scale
  Baseline | 1.00 (0.446) | 0.91 (0.522)
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -0.13 (0.234) | -0.05 (0.114)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -0.26 (0.302) | -0.14 (0.204)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -0.51 (0.382) | -0.32 (0.330)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -0.68 (0.319) | -0.41 (0.428)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -0.83 (0.276) | -0.60 (0.536)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -0.87 (0.311) | -0.70 (0.514)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -0.88 (0.326) | -0.79 (0.582)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -0.88 (0.322) | -0.82 (0.603)

10. Secondary Outcome: Percentage Change From Baseline in F-VASI at Each Post-Baseline Visit
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Percentage change = ([post-Baseline (BL) value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percent change
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -11.69 (20.612) | -6.24 (12.472)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -25.57 (24.957) | -14.62 (20.210)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -54.62 (34.297) | -32.43 (26.031)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -73.31 (27.030) | -40.64 (27.945)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -87.02 (12.247) | -61.31 (28.613)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -89.37 (11.661) | -72.69 (24.815)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -90.44 (11.006) | -80.70 (20.478)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -90.73 (11.002) | -85.55 (15.856)

11. Secondary Outcome: Change From Baseline in T-VASI at Each Post-Baseline Visit
Description: T-VASI was calculated with contributions from 6 body sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each body site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values (range: 0-100; lower scores indicate increased improvement). Change from BL was calculated as the post-BL value minus the BL value.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
scores on a scale
  Baseline | 6.58 (2.163) | 6.87 (2.103)
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -0.40 (0.711) | -0.06 (0.179)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -0.85 (0.865) | -0.17 (0.480)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -1.61 (1.320) | -0.52 (0.710)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -2.47 (1.532) | -0.94 (0.949)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -3.21 (1.686) | -1.73 (1.679)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -3.03 (1.542) | -2.34 (1.746)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -3.42 (1.235) | -2.97 (1.867)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -3.43 (1.219) | -3.46 (2.106)

12. Secondary Outcome: Percentage Change From Baseline in T-VASI at Each Post-Baseline Visit
Description: T-VASI was calculated with contributions from 6 body sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each body site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values (range: 0-100; lower scores indicate increased improvement). Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percent change
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -6.12 (11.217) | -1.02 (3.063)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -15.21 (15.360) | -2.79 (6.833)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -29.76 (24.512) | -7.88 (9.796)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -42.28 (23.530) | -14.82 (15.536)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -57.31 (26.271) | -27.54 (26.386)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -61.19 (28.399) | -35.51 (27.266)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -69.63 (19.748) | -43.76 (27.441)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -69.76 (18.519) | -50.39 (28.689)

13. Secondary Outcome: Change From Baseline in Facial Body Surface Area (F-BSA) at Each Post-Baseline Visit
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of facial surface area
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of facial surface area
  Baseline | 1.12 (0.524) | 0.96 (0.615)
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -0.04 (0.126) | -0.02 (0.088)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -0.08 (0.148) | -0.06 (0.194)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -0.25 (0.246) | -0.17 (0.299)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -0.40 (0.283) | -0.22 (0.378)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -0.63 (0.150) | -0.34 (0.426)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -0.70 (0.167) | -0.44 (0.457)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -0.75 (0.207) | -0.58 (0.577)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -0.77 (0.234) | -0.67 (0.716)

14. Secondary Outcome: Percentage Change From Baseline in F-BSA at Each Post-Baseline Visit
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. The area "Face" did not include surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline (BL) value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percent change
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -4.02 (12.769) | -1.50 (4.345)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -7.25 (13.838) | -4.37 (12.349)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -24.12 (22.508) | -14.83 (19.575)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -39.37 (35.289) | -19.34 (23.332)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -65.36 (25.090) | -34.37 (30.969)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -72.67 (20.378) | -45.42 (31.086)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -77.02 (20.748) | -56.25 (31.498)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -78.06 (20.018) | -60.51 (29.172)

15. Secondary Outcome: Change From Baseline in Total Body Surface Area (T-BSA) at Each Post-Baseline Visit
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of total body surface area
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percentage of total body surface area
  Baseline | 7.00 (2.301) | 7.22 (2.118)
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -0.19 (0.701) | -0.02 (0.200)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -0.48 (0.794) | -0.01 (0.430)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -0.96 (0.952) | -0.17 (0.544)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -1.43 (1.359) | -0.34 (0.659)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -2.14 (1.462) | -0.80 (1.538)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -2.13 (1.556) | -1.12 (1.689)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -2.33 (1.617) | -1.50 (1.988)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -2.37 (1.627) | -1.93 (2.312)

16. Secondary Outcome: Percentage Change From Baseline in T-BSA at Each Post-Baseline Visit
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-BL value minus BL value]/BL value) X 100.
Time Frame: Baseline; up to Week 48
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 20 | 35
percent change
  Week 4: number analyzed (Participants) | 16 | 35
  Week 4 | -2.65 (10.057) | -0.36 (3.374)
  Week 8: number analyzed (Participants) | 14 | 35
  Week 8 | -7.71 (13.609) | -0.24 (6.006)
  Week 12: number analyzed (Participants) | 11 | 35
  Week 12 | -16.92 (17.590) | -2.60 (7.586)
  Week 16: number analyzed (Participants) | 7 | 35
  Week 16 | -23.09 (22.344) | -5.45 (9.946)
  Week 24: number analyzed (Participants) | 7 | 34
  Week 24 | -38.02 (23.485) | -12.50 (21.869)
  Week 32: number analyzed (Participants) | 6 | 32
  Week 32 | -42.86 (28.257) | -16.91 (23.758)
  Week 40: number analyzed (Participants) | 6 | 28
  Week 40 | -46.61 (29.639) | -21.92 (27.234)
  Week 48: number analyzed (Participants) | 6 | 26
  Week 48 | -47.03 (29.370) | -27.30 (30.712)

17. Secondary Outcome: Plasma Concentration of Ruxolitinib at Weeks 4, 12, and 16
Description: The concentration of ruxolitinib in the plasma was assessed.
Time Frame: pre-application at Weeks 4, 12, and 16
Population: Pharmacokinetic (PK)-Evaluable Population: all participants who applied ruxolitinib 1.5% cream at least once and provided at least 1 post-dose blood sample. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanomolar
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB
Number analyzed (Participants) | 16 | 34
nanomolar
  Week 4: number analyzed (Participants) | 16 | 33
  Week 4 | 18.7 (19.0) | 51.1 (45.4)
  Week 12: number analyzed (Participants) | 11 | 33
  Week 12 | 23.3 (23.1) | 53.7 (55.0)
  Week 16: number analyzed (Participants) | 5 | 34
  Week 16 | 49.3 (38.8) | 55.4 (43.9)

ADVERSE EVENTS:
Time Frame: up to approximately 52 weeks
Description: After the 12-week run-in, in which all participants applied ruxolitinib 1.5% cream BID, participants received either ruxolitinib 1.5% cream BID alone or ruxolitinib 1.5% cream BID plus NB-UVB phototherapy for 36 weeks, based on their T-VASI score at Week 12. As pre-specified in the Statistical Analysis Plan, AE data were summarized based on the treatments that the participant received after run-in.
Groups:
- Total: Total
Arm/Group | Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID + NB-UVB | Total
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/35 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/35 | 2/55
Other Adverse Events (participants affected / at risk) | 9/20 | 15/35 | 24/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 1.5% Cream BID (N=20) | Ruxolitinib 1.5% Cream BID + NB-UVB (N=35) | Total (N=55)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 1.5% Cream BID (N=20) | Ruxolitinib 1.5% Cream BID + NB-UVB (N=35) | Total (N=55)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Application site acne (General disorders) | 2 (2) | 4 (4) | 6 (6)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 4 (5)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2)
Scalp haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 3 (4) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT05247489/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT05247489/SAP_001.pdf